CLINICAL TRIAL: NCT06242223
Title: Effects of Multimodal High Intensity Interval Training on Speed, Agility and Performance Level in Cricket Players
Brief Title: Multimodal HIIT in Speed, Agility and Performance Level
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 42667
Record Dates: First submitted 2024-01-28; First posted 2024-02-05 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-01

CONDITIONS: High Intensity Interval Training
Keywords: HIIT; speed; agility; performance level; cricket players; multimodal

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multimodal HIIT (Active Comparator): multimodal HIIT protocol followed by sprinting
  Interventions: Other: Multimodal HIIT
- conventional HIIT (Experimental): Conventional protocol with 4-5 repetitions of 40 seconds maximum running
  Interventions: Other: conventional HIIT

INTERVENTIONS:
Other: Multimodal HIIT — multimodal HIIT protocol followed by sprinting followed by 2 minutes of rest, burpees with 3 minutes rest between sets and push ups 4-5 rep at 80-100% of HR max with a total of 20 minutes exercise per session a day 3 times a week followed by 6 weeks.
  Arms: Multimodal HIIT
Other: conventional HIIT — conve protocol with 4-5 repetitions of 40 seconds maximum running at 80-100% HR max followed by 20 seconds of walking for 20 minutes exercise per session 3 times a week followed by 6 weeks.
  Arms: conventional HIIT

SUMMARY:
The aim of this study is to find out the effect of multimodal high intensity interval training on speed, agility and performance among cricket player.

DETAILED DESCRIPTION:
The literature gap concerns the lack of studies examining the long-term effect of High-Intensity Interval Training (HIIT) on agility performance. Most studies have only examined the acute or short-term effects of HIIT on agility performance, with fewer studies investigating the effect of long-term HIIT interventions on agility performance. Therefore, further research is needed to investigate the efficacy of long-term HIIT interventions in improving agility performance. Additionally, more research is needed to examine the effects of different HIIT protocols on agility performance, as this can help identify the most effective HIIT protocols for improving agility and speed.

Multi-modal high-intensity exercises encompass various workout forms designed to focus on speed, agility, and overall fitness. Research indicates their alignment with the principles of high-intensity interval training (HIIT), highlighting enhanced speed, agility, and metabolic rate improvements.

ELIGIBILITY:
Inclusion Criteria:

It include male and female both, sports specific performance, participants with 18 to 30 years, professional cricket players, willing to follow instructions and athletes who volunteered to participate in the study.

Exclusion Criteria:

It include participants with any associated systemic involvement, any neuro-musculoskeletal problem and with any respiratory and cardiac disease.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-05-08 (Actual); Primary Completion 2024-02-08 (Estimated); Study Completion 2024-02-08 (Estimated)

PRIMARY OUTCOMES:
HIIT | 6 weeks
  HIIT is a type of interval training exercise. It incorporates several rounds that alternate between several minutes of high intensity movements to significantly increase the heart rate to at least 80% of one's maximum heart rate, followed by short periods of lower intensity movements.

SECONDARY OUTCOMES:
speed test | 6 weeks
  sprint distance of 17.68 meters, using the lines on a cricket pitch.
agility t test | 6 weeks
  The T-Test is a simple running test of agility, involving forward, lateral, and backward movements, appropriate to a wide range of sports. purpose: the T-Test is a test of agility for athletes, and includes forward, lateral, and backwards running.
Level of performance scale (LSPS) | 6 weeks
  Performance rating scales are used to assess employee performance in the workplace. They offer a means of gauging job-related abilities, behaviours, and qualifications. Constructing a performance rating system necessitates contemplation of several elements. Total score is 60 and minimum score is 0

CONTACTS AND LOCATIONS:
Overall Officials: sana batool, masters, Principal Investigator — Riphah International University
Locations (1):
- Pakistan Sports Board, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Buchheit M, Laursen PB. High-intensity interval training, solutions to the programming puzzle. Part II: anaerobic energy, neuromuscular load and practical applications. Sports Med. 2013 Oct;43(10):927-54. doi: 10.1007/s40279-013-0066-5. PMID 23832851
- [Background] Ito S. High-intensity interval training for health benefits and care of cardiac diseases - The key to an efficient exercise protocol. World J Cardiol. 2019 Jul 26;11(7):171-188. doi: 10.4330/wjc.v11.i7.171. PMID 31565193
- [Background] Weston M, Weston KL, Prentis JM, Snowden CP. High-intensity interval training (HIT) for effective and time-efficient pre-surgical exercise interventions. Perioper Med (Lond). 2016 Jan 14;5:2. doi: 10.1186/s13741-015-0026-8. eCollection 2016. PMID 26770671
- [Background] Noakes TD, Durandt JJ. Physiological requirements of cricket. J Sports Sci. 2000 Dec;18(12):919-29. doi: 10.1080/026404100446739. PMID 11138982
- [Background] Sharp T, Grandou C, Coutts AJ, Wallace L. The Effects of High-Intensity Multimodal Training in Apparently Healthy Populations: A Systematic Review. Sports Med Open. 2022 Mar 29;8(1):43. doi: 10.1186/s40798-022-00434-x. PMID 35348924